CLINICAL TRIAL: NCT05151523
Title: Long-term Recurrence Rates of Atrial Fibrillation Following New-onset Atrial Fibrillation During ICU Admission
Status: Not yet recruiting | Type: Observational
Sponsor: Katia Orvin (Other)
Responsible Party: Sponsor-Investigator, Katia Orvin, Katia Orvin M.D - director of cardiac intensive care unit, Rabin Medical Center, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Other Study IDs: 0318-21-RMC
Record Dates: First submitted 2021-11-03; First posted 2021-12-09 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; intensive care unit
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Primary Objective of the study is to establish the One-year recurrence rates of atrial fibrillation (AF) following new-onset atrial fibrillation during intensive care unit (ICU) admission.

The Secondary Objective is a composite of death from cardiovascular causes, stroke (either ischemic or hemorrhagic), or hospitalization with worsening of heart failure or recurrent AF.

The prevalence and recurrence rates of AF will be divided into sub-groups based on primary ICU admission diagnosis.

All-cause mortality.

DETAILED DESCRIPTION:
Patients will be screened for atrial fibrillation during hospitalization in the intensive care unit and will be followed until discharge. Once discharged home or to a rehabilitation center, they will be invited to a routine follow-up clinic at RMC cardiology institute 4-6 weeks after hospital discharge. During the clinic visit, patients will be recruited to the study follow-up plan.

The follow-up plan will consist of 3 clinical visits at 4-6 weeks, 6-months and 1 -year after discharge.

The follow-up program will include a comprehensive screening for symptomatic and asymptomatic atrial fibrillation events as following:

Patients will be provided with a home cellular-digital 12-lead ECG transmitter. They will be instructed to conduct routine weekly transmission in order to record asymptomatic events as well as to transmit at any time they suspect an event/feel symptoms (palpitations). Home routine testing will be initiated and guided by a telephone call from a medical monitoring center. A blinded, independent, on-call medical professional team will analyze the received ECG.

A 48-hour Holter ECG will be performed at 6 months and 12 months after ICU discharge

Clinical visits will include 12 leads ECG, physical examination, vital signs, symptoms evaluation for suspected AF events, questioning for hospital admissions, or any other documented AF event. Patients will be asked to perform echocardiography as part of their clinical evaluation. For both the study and control group, documented AF events will be managed according to physician discretion based on clinical practice and guidelines.

Long-term follow-up- 3 years- data regarding recurrent events of AF, hospitalization due to thromboembolic events, and mortality will be evaluated by telephone call or by matching patient identification numbers with the Israeli National Population Register.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU over 24 hours
* Diagnosed with new-onset atrial fibrillation
* The patient survived the index hospitalization and was discharged home/ to a rehabilitation center.

Exclusion Criteria:

• Previously documented atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with new-onset atrial-fibriltion using 30-second telemetry recording or a 12 lead ECG indicating AF during general ICU hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence rates of atrial-fibrillation following new-onset atrial-fibrillation during intensive care unit | One-year
  A positive ECG or Holter test for atrial fibrillation will be regarded as recurrence.

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 3-years
  A composite of death from cardiovascular causes, stroke (either ischemic or hemorrhagic), or hospitalization with worsening of heart failure or recurrent AF.
Recurrence rates of atrial-fibrillation | 3-years
  The prevalence and recurrence rates of atrial-fibrillation divided into sub-groups based on primary ICU admission diagnosis.
All-cause mortality | 3-years
  All-cause mortality will be monitored on clinical flow-up.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boriani G, Fauchier L, Aguinaga L, Beattie JM, Blomstrom Lundqvist C, Cohen A, Dan GA, Genovesi S, Israel C, Joung B, Kalarus Z, Lampert R, Malavasi VL, Mansourati J, Mont L, Potpara T, Thornton A, Lip GYH; ESC Scientific Document Group. European Heart Rhythm Association (EHRA) consensus document on management of arrhythmias and cardiac electronic devices in the critically ill and post-surgery patient, endorsed by Heart Rhythm Society (HRS), Asia Pacific Heart Rhythm Society (APHRS), Cardiac Arrhythmia Society of Southern Africa (CASSA), and Latin American Heart Rhythm Society (LAHRS). Europace. 2019 Jan 1;21(1):7-8. doi: 10.1093/europace/euy110. No abstract available. PMID 29905786
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Result] Kanji S, Williamson DR, Yaghchi BM, Albert M, McIntyre L; Canadian Critical Care Trials Group. Epidemiology and management of atrial fibrillation in medical and noncardiac surgical adult intensive care unit patients. J Crit Care. 2012 Jun;27(3):326.e1-8. doi: 10.1016/j.jcrc.2011.10.011. Epub 2012 Jan 4. PMID 22226423
- [Result] McIntyre WF, Um KJ, Cheung CC, Belley-Cote EP, Dingwall O, Devereaux PJ, Wong JA, Conen D, Whitlock RP, Connolly SJ, Seifer CM, Healey JS. Atrial fibrillation detected initially during acute medical illness: A systematic review. Eur Heart J Acute Cardiovasc Care. 2019 Mar;8(2):130-141. doi: 10.1177/2048872618799748. Epub 2018 Nov 7. PMID 30403364
- [Result] Lubitz SA, Yin X, Rienstra M, Schnabel RB, Walkey AJ, Magnani JW, Rahman F, McManus DD, Tadros TM, Levy D, Vasan RS, Larson MG, Ellinor PT, Benjamin EJ. Long-term outcomes of secondary atrial fibrillation in the community: the Framingham Heart Study. Circulation. 2015 May 12;131(19):1648-55. doi: 10.1161/CIRCULATIONAHA.114.014058. Epub 2015 Mar 13. PMID 25769640
- [Result] Walkey AJ, Hammill BG, Curtis LH, Benjamin EJ. Long-term outcomes following development of new-onset atrial fibrillation during sepsis. Chest. 2014 Nov;146(5):1187-1195. doi: 10.1378/chest.14-0003. PMID 24723004
- [Result] Gialdini G, Nearing K, Bhave PD, Bonuccelli U, Iadecola C, Healey JS, Kamel H. Perioperative atrial fibrillation and the long-term risk of ischemic stroke. JAMA. 2014 Aug 13;312(6):616-22. doi: 10.1001/jama.2014.9143. PMID 25117130